CLINICAL TRIAL: NCT03599440
Title: Evaluation of the Effect of Different Types of Extended Infusion Lines on Pulse Contour-based Measurements Based on the Arterial Pressure Signal
Brief Title: Effect of Extended Infusion Lines on Pulse Contour-based Measurements
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthesist, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: MMS.2018.004
Record Dates: First submitted 2018-06-20; First posted 2018-07-26 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Hemodynamic Instability
Keywords: cardiac output; pulse contour analysis; stroke volume; hemodynamic monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulse contour disturbance: Patients with an arterial catheter and pressure line extensions.
  Interventions: Other: Pressure line extensions

INTERVENTIONS:
Other: Pressure line extensions — Two types of extension lines are connected:
  * Perfusor® line 150cm (polyethylene)
  * conventional arterial extension line

SUMMARY:
Hemodynamic monitoring of the critically-ill patients is increasingly performed using an arterial pulse contour-based cardiac output device such as the proAQT system.

The aim of this study is to evaluate the effect of extending the pressure lines on the arterial pressure wave and the calculated hemodynamic variables when using the proAQT system.

DETAILED DESCRIPTION:
Hemodynamic continuous monitoring of critically-ill patients is increasingly performed with minimally-invasive methods, such as the proAQT sensor (PULSION Medical Systems SE, Munich, Germany).

The proAQT sensor calculates hemodynamic variables such as the cardiac output, stroke volume (variation), pulse-pressure variation and systemic vascular resistance by pulse contour analysis of the arterial pressure waveform using an arterial radial or femoral catheter. This minimal invasive technique, also permits continuous beat-to-beat assessment.

In patients in who an arterial catheter is placed for clinical reasons, the hemodynamic variables are continuously recorded. An extension line is coupled to a 3-way stopcock, connected to the proAQT sensor. In a neutral position of the 3-way stopcock, the pressure wave travels from the pressure sensor through the standard line. By turning the handle of the stopcock the standard line is bypassed and the pressure wave travels through the extended line.

The hemodynamic registration will be as follows:

* two minutes in the neutral position;
* two minutes with one type of extension line
* two minutes in the neutral position
* two minutes with a second type of extension line
* two minutes in neutral position

The arterial pressure curve and all calculated hemodynamic variables are electronically registered.

The influence of two types of extension lines on the accuracy of the calculated hemodynamic variables will be evaluated by comparing the variables measured in neutral position and variables measured with the extended pressure lines. The changes in the calculated variables will be correlated to possible arterial pressure waveform modifications and used to evaluate different algorithms, which might be used to reconstruct the primary pressure wave.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* arterial catheter necessary for clinical reasons

Exclusion Criteria:

* ≥ASA 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients for which arterial pressure measurement is needed.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
relative change in ProAQT-calculated cardiac output after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  relative change (in % of the baseline measurement) in cardiac output following increase in length of the extension line.

SECONDARY OUTCOMES:
change in Area Under the Curve (AUC) of the arterial pressure wave form after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  The relative chane in AUC of the arterial pressure curve (from start systole to dicrotic notch) following increase in length of the extension line.
relative change in ProAQT-calculated SVR after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  relative change (in % of the baseline measurement) in systemic vascular resistance following increase in length of the extension line.
relative change in ProAQT-calculated diastolic blood pressure after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  relative change (in % of the baseline measurement) in diastolic blood pressure following increase in length of the extension line.
relative change in ProAQT-calculated systolic blood pressure after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  relative change (in % of the baseline measurement) in systolic blood pressure following increase in length of the extension line.
relative change in ProAQT-calculated stroke volume variation after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  relative change (in % of the baseline measurement) in stroke volume variation following increase in length of the extension line.
relative change in ProAQT-calculated pulse pressure variation after placement of extension lines. | one minute of measurement after changing the length of the extension line.
  relative change (in % of the baseline measurement) in pulse pressure variation following increase in length of the extension line.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Kalmar, MD, PhD, MSc, Principal Investigator — Maria Middelares Hospital
Locations (1):
- AZ Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No